CLINICAL TRIAL: NCT05695157
Title: Clinical Performance and Safety of Suture-TOOL for Abdominal Wound Closure in Men and Women Patients Undergoing Elective Open Abdominal Surgery
Brief Title: Clinical Performance and Safety of Suture-TOOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suturion AB (Industry)
Collaborators: Helsingborgs Hospital (Other); Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRO-21-149; CIV-22-09-040607 (Other: Swedish Medical Products Agency); SUT 001 (Other: Suturion AB)
Record Dates: First submitted 2023-01-09; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Laparotomy; Incisional Hernia; Wound Infection; Closure Technique
MeSH Terms: conditions — Incisional Hernia; Wound Infection

STUDY DESIGN:
Intervention Model Description: Single arm prospective interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Closure of the abdomen after laparotomy with Suture-TOOL.
  Interventions: Device: Suture-TOOL

INTERVENTIONS:
Device: Suture-TOOL — Suture device for fast and standardized closure of the abdominal fascia

SUMMARY:
The goal of this single arm intervention study is to investigate the safety and performance of a suturing device for closure of the midline incision after open abdominal surgery. The study population consists of 38 patients selected for open abdominal procedures for malignant and benign colorectal disease.

The main question it aims to answer is:

• If the device facilitates a Suture-Length to Wound-Length (SL/WL) ratio of 4:1

Participants laparotomy wound will be closed with the device at the end of the operation and closure related data as closure time and SL/WL ratio will be calculated. The wound will be assessed for infection during the postoperative stay and the chart will be reviewed for wound dehiscence and wound infection.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the investigation
2. Sex, age: male and female patients, ≥ 18 years old
3. Surgery: elective open abdominal surgery for benign or malignant colorectal disease through midline incision.

   Anticipated incision length ≥ 12 cm
4. Body Mass Index (BMI): 18 - 40 kg/m2 inclusive
5. Full comprehension: ability to comprehend the full nature and purpose of the investigation, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire investigation.

Exclusion Criteria:

1. Abdominal Surgery: previous abdominal surgery involving the midline
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the investigation according to the Investigator's opinion; existing midline hernia, cutaneous infection, fistula, psoriasis of abdominal skin; morbidly obese patients
3. Pre-operative findings: any pre-operative findings identified by the surgeon/Investigator that may preclude the conduct of the investigation procedures
4. Allergy: history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers could affect the outcome of the investigation
5. Diseases: known or identified at surgery disseminated cancer disease; collagen diseases and immune deficiency disorders, according to the Investigator's opinion. Significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that according to the Investigator's opinion may interfere with the aim of the investigation
6. Life expectancy: life expectancy less than 1 year
7. Medications: any medication that could interfere with the investigation procedures or investigation outcome, according to the Investigator's opinion. Hormonal contraceptives for women are allowed
8. Pregnancy and lactation: positive pregnancy test at screening (if applicable); pregnant or breastfeeding women
9. Vulnerable subjects: Individuals unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced because of a compromised position, expectation of benefits or fear of retaliatory response (ISO 14155:2020 §3.55) will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Suture length/Wound length (SL/WL) ratio ≥ 4 | Measured during laparotomy closure.
  SL/WL-ratio of patients laparotomy closures will be calculated by measuring (centimeter) and dividing the length of used suture with the length of the laparotomy wound.

SECONDARY OUTCOMES:
Stitch count | Measured during laparotomy closure
  Number of stitches used for laparotomy closure
Numbers of sutures used | Counted during laparotomy closure
Incision closure time | Measured during laparotomy closure
  Time (seconds) from first to last knot during laparotomy closure
Surgeons´ comfort with device during closure | After laparotomy closure
  VAS assessment
Surgeons´ satisfaction with final closure result | After laparotomy closure
  VAS assessment

OTHER OUTCOMES:
Incision not following the midline (exposure of rectus muscle) | During the whole study period of up to 8 months
  Assessment of midline incision
Thickness of subcutaneous fat | During the whole study period of up to 8 months
  Measurement of subcutaneous fat (millimeter)
Glove punctures | During the whole study period of up to 8 months
  Standardized assessment of puncture holes
Re-operation(s) number | 45 days after surgery
  Chart review
Reasons for unscheduled post-surgery visits | 45 days after surgery
  Chart review
Type of adverse effects | During the whole study period of up to 8 months
  All adverse effects derived by spontaneous, unsolicited reports of the subjects or users/handlers, by observation and by routine open questioning will be collected and reported.
Type of adverse device effects | During the whole study period of up to 8 months
  Identification of adverse device effects
Type of device deficiencies | During the whole study period of up to 8 months
  Identification of device deficiences
Reasons for device replacement during surgery | During the whole study period of up to 8 months
  Identification during study period
Patients with wound infections | 45 days after surgery
  Wound infection postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Edelhamre, MD Phd, Principal Investigator — Region Skåne
Locations (1):
- Helsingborgs Hospital, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Borner G, Montgomery A. Suture-Tool: A Mechanical Needle Driver for Standardized Wound Closure. World J Surg. 2020 Jan;44(1):95-99. doi: 10.1007/s00268-019-05179-5. PMID 31549201
- [Result] Borner G, Edelhamre M, Rogmark P, Montgomery A. Suture-TOOL: A suturing device for swift and standardized abdominal aponeurosis closure. Surg Pract Sci. 2022 Oct 5;11:100137. doi: 10.1016/j.sipas.2022.100137. eCollection 2022 Dec. PMID 39845163